CLINICAL TRIAL: NCT02212314
Title: Developing Treatments to Improve Psychosocial Functioning in Children With Williams Syndrome Part 1: Response Inhibition Training for Children With Williams Syndrome
Brief Title: Response Inhibition Training for Children With Williams Syndrome
Acronym: WSRIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Milwaukee (Other)
Responsible Party: Principal Investigator, Bonita P Klein-Tasman, Professor, University of Wisconsin, Milwaukee
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 14.351
Record Dates: First submitted 2014-08-06; First posted 2014-08-08 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Williams Syndrome
Keywords: Response Inhibition, Williams Syndrome
MeSH Terms: conditions — Williams Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Response Inhibition Training (Experimental): Treatment group will receive immediate treatment after pre-test.
  Interventions: Behavioral: Response Inhibition Training
- Waitlist Crossover (No Intervention): Waitlist group will not receive intervention while treatment group is active, but waitlist group will be offered treatment after post-test is completed.

INTERVENTIONS:
Behavioral: Response Inhibition Training — Computerized response inhibition training will be delivered via the Internet for 10 individual sessions.
  Arms: Response Inhibition Training

SUMMARY:
The investigators will conduct a pilot study investigating the effectiveness of a computerized response inhibition training program at reducing the response inhibition difficulties often seen in children with Williams syndrome ages 10-17. The investigators hypothesize that after completing the training program, children with Williams syndrome will show improvement on computerized measures of response inhibition and on parent measures of impulsivity.

DETAILED DESCRIPTION:
Behavioral characteristics of individuals with Williams syndrome include eagerness to approach and interact with others (including strangers), repeated questions especially about upcoming events, and difficulties with attention, impulsivity, and inhibition. There is very little systematic research about the kinds of interventions that are most useful for children with Williams syndrome to support optimal psychosocial functioning, and of the effectiveness of such interventions. We will conduct a pilot study of a potential intervention to address the response inhibition difficulties associated with Williams syndrome. The investigators will examine the utility of an online, web-based computerized cognitive retraining program aimed at addressing impulsivity and inhibition difficulties in 20 children, ages 10-17, with WS. The engaging training program has shown some utility in other populations, including children with tic disorders and trichotillomania. The investigators will examine the acceptability and feasibility of the treatment approach, as well as its impact on performance on experimental measures of impulsivity and on everyday psychosocial functioning as rated by parents; this study will consist of a small-scale pilot Randomized Clinical Trial with wait list. Through this novel work, we hope to develop and tune this approach for optimal outcomes and to demonstrate the promise of this intervention to address common challenges of people with Williams syndrome in the area of inhibition.

ELIGIBILITY:
Inclusion Criteria:

* Williams syndrome (diagnosed with genetic testing)
* Ages 10-17
* First language and main language spoken in the home is English
* Possess computer in the home that has internet access, and a second electronic device with access to Skype (e.g., smartphone, ipad, additional computer, ipod touch)

Exclusion Criteria:

* First language and main language spoken in the home is NOT English (because study measures and instructions are all in English)
* No computer in the home with internet access (because the study is being conducted via the internet)
* Comorbid severe illnesses or major surgery within the past 6 months
* Four or more previous sessions of inhibition training

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2014-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Cognitive Inhibition Tasks | 5-7 weeks and 3 months
  Three measures of response inhibition that were administered to children at pre-test will be administered after the 5-7-week training and again at a 3-month follow-up. Measures include computer-administered Motor Stroop task, Stop Signal task, and Go/No-Go Task.

SECONDARY OUTCOMES:
Conners-3 | 5-7 weeks and 3 months
  The Conners-3 will be administered to parents at post-intervention and again at follow-up to assess changes in attention and impulsivity.
Emotion Regulation Checklist | 5-7 weeks and 3 months
  The Emotion Regulation Checklist will be administered to parents at post-intervention and follow-up to assess changes in the child's ability to regulate emotions.
Positive and Negative Affect Scale | 5-7 weeks and 3 months
  The PANAS will be administered to parents at post-intervention and follow-up to assess changes in child positive and negative affect.
Question-Asking Questionnaire | 5-7 weeks and 3 months
  The QAQ will be administered to parents at post-intervention and follow-up to assess changes in amount and frequency of child anticipatory question asking.
Spence Children's Anxiety Scale | 5-7 weeks, 3 months
  The SCAS will be administered to parents at post-intervention and follow-up to assess changes in child anxieties.
MINI Kid 6.0 Parent Version | 5-7 weeks and 3 months
  The MINI Kid 6.0 Parent will be administered to parents at post-intervention and follow-up to assess changes in those areas endorsed at pre-intervention.

OTHER OUTCOMES:
Treatment Acceptability Questionnaire | 5-7 weeks
  Questionnaire about study acceptability will be administered at post test after the 5-7 week training.
Treatment Evaluation Inventory | 5-7 weeks
  Questionnaire evaluating treatment will be administered at post test after the 5-7 week training.

CONTACTS AND LOCATIONS:
Overall Officials: Bonita P Klein-Tasman, Ph.D., Principal Investigator — University of Wisconsin, Milwaukee
Locations (1):
- University of Wisconsin-Milwaukee Child Neurodevelopment Research Lab, Milwaukee, Wisconsin, United States